CLINICAL TRIAL: NCT00367575
Title: An Internet-based Intervention for Problem Drinking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 053/2005
Record Dates: First submitted 2006-08-21; First posted 2006-08-23 (Estimated); Last update posted 2010-08-16 (Estimated); Status verified 2010-08

CONDITIONS: Alcoholism
Keywords: alcoholism; drinking; randomized; internet personalized alcohol feedback
MeSH Terms: conditions — Alcoholism | interventions — Ethanol

INTERVENTIONS:
Procedure: Internet personalized alcohol feedback (PAF)

SUMMARY:
The main aim of this randomized controlled trial is to evaluate the efficacy of an Internet-delivered self-help intervention for problem drinkers in the general population.

Adult problem drinkers with home access to the Internet will be recruited from the CAMH Monitor. Subjects will be randomly assigned to receive a website address where they can obtain personalized feedback about their drinking, or to a no intervention control group.

Three-month and six-month follow-up surveys will be conducted by mail to assess drinking over the following three month periods. Collaterals will be requested and interviewed after the six-month follow-up. Subjects will be paid $40.00 and collaterals will be paid $20.00 for their participation. Drinking at three- and six-months will be compared between the groups. Subjects in the control group will be provided with the website address following the six-month follow-up.

DETAILED DESCRIPTION:
Self-change interventions have great potential to aid the many problem drinkers who do not seek formal treatment. Because self-change interventions circumvent some of the barriers associated with traditional treatment services, they may help reduce the harm associated with alcohol abuse among untreated individuals, whose number far exceeds that of the minority who ever access formal alcohol treatment programs. Self-change/self-help materials have the added advantage of being relatively inexpensive, increasing their potential for wide distribution and attendant public health impact. The Internet is one promising route for distributing such materials to a large segment of the population. Three-quarters of Canadians and Americans use the Internet, including a large number who seek health-related information on line. Drinking self-change websites abound on the Internet, but because none has been scientifically evaluated it is unknown whether such sites do more good than harm.

By being the first large scale, controlled evaluation, this project intends to advance the science of Internet-mediated intervention as well as provide valuable public health information on the effectiveness of Internet-delivered self-change materials. Specifically, the major objective of this project is to conduct a randomized controlled evaluation of the impact of an Internet-based self-help intervention for problem drinkers in the general population.

Participants will be recruited through the ongoing general population survey - the CAMH Monitor (N = 170 after attrition), and will be randomly assigned to be sent a World Wide Web page Internet address and password for the personalized alcohol feedback program or to a no intervention control group. Three and six-month drinking outcomes will be compared between experimental conditions using structural equation modeling.

The primary hypothesis is that respondents in the Internet personalized alcohol feedback condition will display significantly improved drinking outcomes at three and six-month follow-ups as compared to respondents in the no intervention control condition. Secondary hypotheses will address the mediating or moderating role of perceived drinking norms, perceived risk and the problem drinker's social reasons for drinking.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* have home access to the Internet
* interested in receiving a computerized assessment of their drinking
* have a score of 8 or higher on the AUDIT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 359 (Estimated)
Dates: Start 2006-09; Study Completion 2009-09

PRIMARY OUTCOMES:
frequency of consumption
drinks per occasion
number of drinks in a typical week
frequency of 5+ consumption
highest number of drinks on one occasion.

CONTACTS AND LOCATIONS:
Overall Officials: John A Cunningham, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (3):
- Stanford University School of Medicine, Stanford, California, United States
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - Centre for Addiction and Mental Health, Toronto, Ontario

REFERENCES:
- [Derived] Cunningham JA, Wild TC, Cordingley J, Van Mierlo T, Humphreys K. Twelve-month follow-up results from a randomized controlled trial of a brief personalized feedback intervention for problem drinkers. Alcohol Alcohol. 2010 May-Jun;45(3):258-62. doi: 10.1093/alcalc/agq009. Epub 2010 Feb 10. PMID 20150170